CLINICAL TRIAL: NCT04243096
Title: Wearable Sensor-based Outcomes Following Physical Therapy in Knee Osteoarthritis: A Feasibility Study (WESENS-OA)
Brief Title: Wearable Sensors in Knee OA
Acronym: WESENS-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Boston University (Other); Pfizer (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Deepak Kumar, Assistant Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5540E
Record Dates: First submitted 2020-01-14; First posted 2020-01-28 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
Keywords: physical therapy; wearable sensors; gait; pain sensitization; physical activity
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-arm interventional study
Masking Description: Since this is a single-arm study, no masking is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise-based Physical Therapy (Experimental): 12 week in-person exercise-based physical therapy
  Interventions: Behavioral: Exercise-based Physical Therapy

INTERVENTIONS:
Behavioral: Exercise-based Physical Therapy — Exercises for pain modulation, strengthening, and neuromuscular control
  Other Names: Exercise

SUMMARY:
This is a single-arm clinical trial to investigate the outcome of exercise-based physical therapy in people with knee osteoarthritis through the use of wearable sensors.

DETAILED DESCRIPTION:
This is a longitudinal, single arm, 19-week study to investigate the utility of digital assessments to measure the efficacy of exercise-based physical therapy (PT) for reducing pain and improving function in people with knee osteoarthritis (OA).

A total of 60 participants will be included. Participants will receive a supervised exercise-based PT for 12 weeks and will undergo multiple assessments of strength, balance, gait and joint movement while being monitored with a motion capture system and wrist and lumbar wearable sensors. Additionally, participants' activities will be monitored in the real world with the same wrist and lumbar wearable sensors. After completion of the PT program, participants will be monitored for an additional 6-week period to measure persistence of treatment effect. During that time, they will continue to follow an exercise program at home.

The primary objective will be to measure the effect of exercise-based PT on functional performance and pain reduction using both patient reported outcomes questionnaires (PROs) and digital metrics obtained from the laboratory assessments and wearable sensors worn in the real world. Pain phenotyping questionnaires and quantitative sensory testing assessments will also be used to evaluate the effect of specific pain phenotypes in treatment response.

A substudy will be undertaken to assess reproducibility of sensor-based measures during physical performance testing across at-home and in-lab implementation, as well as, reproducibility of these measures over repeated at-home implementation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years of age
* A confirmed clinical diagnosis of osteoarthritis of the knee based on American College of Rheumatology criteria (confirmed by the participant's physician).
* Score ≥ 3 on weight-bearing questions from the Knee injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale in the index knee
* BMI ≤ 40 kg/m2
* Able to walk without assisted devices (eg. cane or walker) for at least 20 minutes
* Can speak and understand English
* Available for the study duration

Exclusion Criteria:

* Contraindication to exercise
* Other pain in lower back or legs that is greater than knee pain
* Currently receiving chemotherapy or radiation therapy for cancer except non-melanoma skin cancer
* History of other disease that may involve the index joint including inflammatory joint disease such as rheumatoid arthritis, seronegative spondyloarthropathy (eg, ankylosing spondylitis, psoriatic arthritis, inflammatory bowel disease related arthropathy), crystalline disease (eg, gout or pseudogout), lupus erythematosus, knee joint infections, Paget's disease affecting the knee, or knee joint tumors.
* Any knee surgery in the previous 6 months
* Previous knee osteotomy, uni-compartmental replacement, or total knee replacement in either knee
* Joint replacement in either hip or ankle
* Planned major treatment for knee OA (e.g., surgery, injections, physical therapy) during the study period
* Planned major surgery in the next 6 months
* Corticosteroid or hyaluronic acid injections in either knee in the previous 3 months
* Neurological conditions that impacts motor functioning, for e.g., stroke, Parkinson's disease, Alzheimer's disease, Multiple Sclerosis, diabetic neuropathy, etc.
* Pregnant
* Received physical therapy for knee OA within past 6 months
* Known or suspected non-compliance, drug or alcohol abuse
* Participation in another clinical trial for treatment of any joint or muscle pain
* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigators.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kumar, PT, PhD, Principal Investigator — Boston University; Tuhina Neogi, MD, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publication(s), after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following publication(s).
Access Criteria: Data will only be shared for individual participant data meta-analyses. Data will be shared with investigators who propose a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Lee S, Neogi T, Costello KE, Senderling B, Stefanik JJ, Frey-Law L, Kumar D. Association of mechanical temporal summation of pain with muscle co-contraction during walking in people with knee osteoarthritis. Clin Biomech (Bristol). 2023 Dec;110:106105. doi: 10.1016/j.clinbiomech.2023.106105. Epub 2023 Sep 22. PMID 37778085
- [Derived] Rose MJ, Neogi T, Friscia B, Torabian KA, LaValley MP, Gheller M, Adamowicz L, Georgiev P, Viktrup L, Demanuele C, Wacnik PW, Kumar D. Reliability of Wearable Sensors for Assessing Gait and Chair Stand Function at Home in People With Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2023 Sep;75(9):1939-1948. doi: 10.1002/acr.25096. Epub 2023 Mar 7. PMID 36734316

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise-based Physical Therapy
Started | 62
Completed | 58
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 50
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 60
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.0 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Sensor Derived Cadence
Description: number of steps/min during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: steps/min
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
steps/min | 4.62 [2.60 to 6.64]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.62, 95% CI 2-sided [2.60 to 6.64]

2. Primary Outcome: Sensor Derived Stride Duration
Description: duration of one stride during gait (sec) during the clinic-based 28-meter walk test
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: second
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
second | -0.04 [-0.06 to -0.02]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.06 to -0.02]

3. Primary Outcome: Sensor Derived Step Duration
Description: duration of one step during gait (sec) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: second
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
second | -0.02 [-0.03 to -0.01]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.03 to -0.01]

4. Primary Outcome: Sensor Derived Stance Time
Description: Duration of stance phase (i.e., duration of time the foot is in contact with the ground in a step) during gait (sec) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: second
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
second | -0.03 [-0.04 to -0.02]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.04 to -0.02]

5. Primary Outcome: Sensor Derived Total Double Support Time
Description: time when both feet are on the ground in one gait cycle (sec) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
seconds | -0.01 [-0.01 to 0.00]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.01 to 0.00]

6. Primary Outcome: Sensor Derived Swing Time
Description: duration of swing phase during gait (sec) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
seconds | -0.01 [-0.02 to -0.01]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p = 0.0013, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.02 to -0.01]

7. Primary Outcome: Sensor Derived Single Limb Support Time
Description: time when one foot is on the ground in one gait cycle (sec) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
seconds | -0.02 [-0.02 to -0.01]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.02 to -0.01]

8. Primary Outcome: Sensor Derived Step Length
Description: length of a step during gait (m) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
meters | 0.03 [0.02 to 0.04]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [0.02 to 0.04]

9. Primary Outcome: Sensor Derived Gait Speed
Description: walking speed (m/s) during the clinic-based 28-meter walk test from lower back sensor
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 56
m/s | 0.09 [0.06 to 0.13]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.06 to 0.13]

10. Primary Outcome: Sensor Derived Duration of Sit to Stand
Description: time taken to complete a chair stand (sec) from lower back sensor
Time Frame: Change from baseline to 12 weeks
Population: these data were only available from a few participants due to issues with the algorithm
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 6
seconds | 0.20 [-0.41 to 0.80]

11. Primary Outcome: Sensor Derived Sit to Stand Acceleration
Description: peak acceleration during chair stand (m/s^2) from lower back sensor
Time Frame: Change from baseline to 12 weeks
Population: these data were only available from a few participants due to issues with the algorithm
Measure: Mean (95% Confidence Interval); unit: meters per second squared
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 6
meters per second squared | 0.10 [-1.62 to 1.81]

12. Primary Outcome: Sensor Derived Sit to Stand Deceleration
Description: peak deceleration during chair stand (m/s^2) from lower back sensor
Time Frame: Change from baseline to 12 weeks
Population: these data were only available from a few participants due to issues with the algorithm
Measure: Mean (95% Confidence Interval); unit: meters per second squared
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 6
meters per second squared | -0.33 [-2.94 to 2.27]

13. Secondary Outcome: Physical Function (KOOS ADL)
Description: Knee injury and Osteoarthritis Outcome Scale ADL Score (0-100, higher score indicate better outcome)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 55
score on a scale | 9.96 [6.60 to 13.31]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 9.96, 95% CI 2-sided [6.60 to 13.31]

14. Secondary Outcome: Knee Pain (KOOS Pain)
Description: Knee injury and Osteoarthritis Outcome Scale Pain Score (0-100, higher score indicate better outcome)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 55
score on a scale | 13.07 [9.65 to 16.48]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; adjusted for age, sex, BMI, and presence of comorbidities; Mean Difference (Final Values) = 13.07, 95% CI 2-sided [9.65 to 16.48] — Change from baseline to week 12

15. Secondary Outcome: Moderate to Vigorous Physical Activity (MVPA)
Description: time spent in moderate and vigorous intensity activity per day extracted from a wrist worn sensor (GT9X Link)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 53
minutes | -17.5 [-39.7 to 4.61]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p = 0.1196, Mixed Models Analysis; Median Difference (Final Values) = -17.5, 95% CI 2-sided [-39.7 to 4.61]

16. Secondary Outcome: Time Taken to Complete 28-meter Walk Test
Description: time taken to complete 28-meter walk test (s) from stopwatch during the clinic-based 28-meter walk test
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: second
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 58
second | -3.23 [-4.33 to -2.12]

17. Secondary Outcome: First Peak of Knee Index
Description: Knee loading index for study knee during walking at self-selected pace from 3D motion capture (%Bodyweight*height)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: %Newton*meter
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 40
%Newton*meter | 0.11 [-0.04 to 0.25]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.04 to 0.25]

18. Secondary Outcome: Knee Co-contraction
Description: Peak medial quadriceps-medial hamstrings co-contraction during loading response during walking at self-selected pace. Higher values reflect greater co-activation of these muscles.
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 40
arbitrary units | -1.83 [-5.76 to 2.09]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.83, 95% CI 2-sided [-5.76 to 2.09]

19. Secondary Outcome: Knee Frontal Plane Excursion
Description: abduction-adduction range during stance phase of gait measured using 3D motion capture (degrees)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: Degrees
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 58
Degrees | -0.15 [-0.46 to 0.16]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.46 to 0.16]

20. Secondary Outcome: Knee Sagittal Plane Excursion
Description: flexion-extension range for study knee during stance phase of gait measured during walking at self-selected pace using 3D motion capture (degrees)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: degree
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 58
degree | -1.15 [-2.22 to -0.08]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-2.22 to -0.08]

21. Secondary Outcome: Trunk Angle
Description: peak trunk forward flexion angle during sit-to-stand measured using 3D motion capture (degrees)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: degree
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 55
degree | -0.08 [-3.37 to 3.22]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-3.37 to 3.22]

22. Secondary Outcome: Global Assessment
Description: Patient Global Assessment of OA (PGA-OA) (range 0-100, higher score indicates better outcome)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 54
score on a scale | 6.21 [1.31 to 11.11]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p = 0.0134, Mixed Models Analysis; Mean Difference (Final Values) = 6.21, 95% CI 2-sided [1.31 to 11.11]

23. Secondary Outcome: Step Up Test
Description: number of step ups completed in 15 seconds
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: repetitions
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 58
repetitions | 1.75 [1.16 to 2.34]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = 1.75, 95% CI 2-sided [1.16 to 2.34]

24. Secondary Outcome: Stair Climbing Test (SCT)
Description: Time taken to go up and down a flight of stairs (sec)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 57
seconds | -1.19 [-1.97 to -0.41]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p = 0.0030, Mixed Models Analysis; Median Difference (Final Values) = -1.19, 95% CI 2-sided [-1.97 to -0.41]

25. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: Short Physical Performance Battery total score. This is a functional test where several different activities (e.g., balance, walking, getting up from a chair) are performed and scored by the examiner. The total score is the sum of scores across all of the activities. Range is 0-12. Higher scores reflect better physical function.
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 58
score on a scale | 0.45 [0.23 to 0.67]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.23 to 0.67]

26. Secondary Outcome: 6-minute Walk Test (6MWT)
Description: distance covered walking in 6 minutes (m)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 58
meters | 35.18 [18.70 to 51.67]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 35.18, 95% CI 2-sided [18.70 to 51.67]

27. Secondary Outcome: 5-time Sit to Stand (5STS)
Description: time taken to complete 5 chair stands (sec)
Time Frame: Change from baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Exercise-based Physical Therapy
Number analyzed (Participants) | 57
seconds | -1.98 [-2.57 to -1.39]
Statistical Analysis 1: Comparison: Exercise-based Physical Therapy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.57 to -1.39]

28. Other Pre Specified Outcome: Number of Sit to Stand
Description: number of chair stands per day measured using lumbar sensor
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Gait Bouts
Description: number of gait bouts per day measured using lumbar sensor
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Total Sleep Time
Description: total sleep time per day measured using wrist-worn sensor (minutes)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Sleep Interference
Description: Daily Sleep Interference Scale (DSIS) (0-10 numeric rating scale, higher number indicates greater interference in sleep due to pain)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Peak Extensor Isometric Torque
Description: peak extensor muscle torque from isometric strength testing (Nm/kg)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Pressure Pain Threshold (PPT)
Description: pressure at which pain is initially felt (kg/m2)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Temporal Summation (TS)
Description: presence of wind up phenomenon in response to multiple pressure stimuli (yes/no)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Conditioned Pain Modulation (CPM)
Description: reduction in pain sensitivity with application of second pain stimulus (yes/no)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Knee Pain
Description: Numeric rating scale for pain (0-10, higher score indicates worse pain)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Knee Pain During Nominated Activity
Description: Numeric rating scale for pain during nominated activity (0-10, higher score indicates worse pain)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Symptoms - KOOS Symptoms
Description: Knee injury and osteoarthritis outcome score Symptoms scale (0-100, higher scores indicates better outcome)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

39. Other Pre Specified Outcome: QOL - KOOS QOL
Description: Knee injury and osteoarthritis outcome score quality of life scale (0-100, higher scores indicates better outcome)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

40. Other Pre Specified Outcome: S/R - KOOS S/R
Description: Knee injury and osteoarthritis outcome score sports/recreation scale (0-100, higher scores indicates better outcome)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Depressive Symptoms
Description: Center for Epidemiologic Studies Depression Scale (range 0-60, higher score indicate more depressive symptoms)
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Number of Painful Joints
Description: number of painful joints in the body
Time Frame: Change from baseline to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 10months
Arm/Group | Exercise-based Physical Therapy
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise-based Physical Therapy (N=60)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Spinal Tumor (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise-based Physical Therapy (N=60)
Skin Irritation (Skin and subcutaneous tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
All sensor-based results are preliminary. Further optimization of the algorithm is underway.

Sensor-based measures for sit-to-stand were only available from a few participants and hence those data should be interpreted with caution.

The serious adverse events were unrelated to the study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04243096/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04243096/SAP_001.pdf